CLINICAL TRIAL: NCT00380536
Title: Adapting a Medical Self-Management Program for a Community Mental Health Center
Brief Title: Medical Self-Management for Improving Health Behavior Among Individuals in Community Mental Health Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Benjamin Druss, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00047631; R34MH078583 (NIH); DAHBR 96-BHB
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Disease; Mental Illness
Keywords: Peer-led Education
MeSH Terms: conditions — Chronic Disease; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will participate in peer-led medical illness self-management group sessions.
  Interventions: Behavioral: Peer-Led Health Education Class
- 2 (No Intervention): Participants will receive treatment as usual.

INTERVENTIONS:
Behavioral: Peer-Led Health Education Class — Participants will participate in group sessions once a week for 6 weeks. Sessions will focus on medical self-management, healthy behaviors, and effective use of the general medical system.
  Arms: 1

SUMMARY:
This study will evaluate the effectiveness of a medical illness self-management program in improving the health and health behavior of people who are receiving care at a community mental health center.

DETAILED DESCRIPTION:
People with serious mental disorders tend to have shorter life expectancies and elevated rates of unhealthy behaviors and chronic illnesses. Peer-led medical illness self-management programs have been shown to be effective in improving the health and health behaviors of people with chronic medical conditions. This type of intervention, however, has yet to be systematically tested in individuals with mental disorders. Community mental health centers provide care to many people of low socioeconomic status who lack medical insurance. This study will evaluate the effectiveness of a medical illness self-management program in improving the health and health behaviors of people who are receiving care at a community mental health center.

Participants in this study will be randomly assigned to either partake in peer-led medical illness self-management group sessions or receive care as usual. Participants assigned to care as usual will continue to receive any services they would have otherwise been offered, but will not receive any additional services through the study. Participants assigned to the medical illness self-management program will attend group sessions once a week for 6 weeks. Sessions will focus on medical self-management, healthy behaviors, and effective use of the general medical system.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving treatment at Dekalb Community Service Board
* Chronic disease

Exclusion Criteria:

* History of more than two psychiatric or medical hospitalizations within the year prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Patient activation | Measured at Months 6 and 12

SECONDARY OUTCOMES:
Health-related quality of life | Measured at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Druss, MD, MPH, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Winn Way Mental Health Center, Decatur, Georgia
  - Clifton Springs Mental Health Center, Decatur, Georgia